CLINICAL TRIAL: NCT01423669
Title: The Hong Kong Morbidity Survey 2010 Part 3: Epidemiology Study of Psychosis Disorder and Sub-clinical Psychotic Experiences
Brief Title: Epidemiology Study of Psychosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other); Kowloon Hospital, Hong Kong (Other); Castle Peak Hospital (Other Government); North District Hospital, Hong Kong (Unknown); Shatin Hospital (Other); Tai Po Hospital (Other Government); Kwai Chung Hospital (Other); Prince of Wales Hospital, Shatin, Hong Kong (Other)
Responsible Party: Dr May Mei-ling LAM, The University of Hong Kong
Other Study IDs: Epi-2010
Record Dates: First submitted 2011-08-10; First posted 2011-08-26 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Psychotic Disorders
Keywords: Psychotic Disorders
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Community dwelling adult population

SUMMARY:
Purpose Psychotic disorders (including schizophrenia) are complex neurobehaviour disorders influenced by genetic, neurodevelopmental, neurochemical, as well as psychosocial factors. Despite significant progresses in pharmacotherapy, the disorder often results in long-term disability (ranked globally amongst the top ten leading causes of disability-adjusted life years, DALYS), often associated with extensive cost, burden, morbidity and mortality.

Objective / hypothesis The study aims to (1) measure the prevalence of psychotic symptoms in the Hong Kong population; (2) explore associated risk and protective factors for the expression of psychotic symptoms; (3) characterize the functional disability in people with psychotic symptoms; and (4) study the determinant of clinical presentation or non-presentation in people with psychotic symptoms.

Design, subjects and study instrument The survey will be conducted with a two-phase design. The first phase interviews will include approximately 5,000 subjects with structured assessments serving diagnostic criteria for CMD, screening instruments for psychotic disorder, substance misuse and suicidal behaviours, functioning, service use and demographics. The second phase comprises of clinician interviews for psychotic disorder and "at risk mental state" and other variables including neurocognitive, help seeking, stigma and well-being.

Analysis Prevalence estimates will be weighted, expressed as rates and confidence intervals. Comorbidity will be estimated using Latent Class Analysis (LCA) Logistic regression will be used to identify significant factors associated with mental disorders.

DETAILED DESCRIPTION:
Psychotic disorders (including schizophrenia) are complex neurobehaviour disorders influenced by genetic, neurodevelopmental, neurochemical, as well as psychosocial factors. Amongst these risk factors, recent findings have highlighted the roles of immigration, urban upbringing, high paternal age, psychoactive substance abuse, as well as stressful early experiences. Despite significant progresses in pharmacotherapy, the disorder often result in long-term disability ranked globally amongst the top ten leading causes of disability-adjusted life years (DALYS, WHO). The World health Organization concludes that the burden and human suffering associated with psychosis is extensive and results in high service and societal costs. Identification and treatment of psychotic disorders (sometimes referred to as Severe Mental Illness, or SMI) is a priority in most mental health services worldwide. However such efforts are challenging because of the help-seeking is severely compromised by reluctance, stigmatization, lack of knowledge, and poor accessibility. This has resulted in long delays before treatment, as well as lack of information about the community prevalence, and associated disability and risk factors for psychosis (ref DUP paper). Availability of these data for Hong Kong will facilitate service planning, early detection and intervention efforts, as well as the consideration of population level preventative strategies.

Availability data suggest that the prevalence of psychosis in the community is substantially higher (5.5-28%, vanos 09) than the prevalence of treated disorder (1-3.5%, vanos09 ), raising important questions about the what determines whether and when psychotic disorders are intercepted in a particular service setting. It is vital to also to obtain information about the untreated cases, in terms of risk factors and protective factors, disability, as well as obstacles to help-seeking.

Community level data for psychotic disorders in Hong Kong is sparse and there has been no territory-wide population-level epidemiology. The Hong Kong population has several distinctive features which are of particular scientific interest and public health concern in relation to psychosis. Although the overall prevalence of substance abuse is low, there is disproportionate use of ketamine in Hong Kong, which interferes with glutaminergic neurotransmission. The relationship between ketamine use and risk for psychosis is of aetiological and clinical interest. In addition, the unique societal context of Hong Kong has resulted in a high proportion of immigrants from China. Moreover, a cohort of people with relatively high paternal age is entering the risk period of developing psychotic disorders (resulting from older man from Hong Kong and younger women from neighbouring parts of China in the previous decades).

Previous relevant study included a district survey, which was more than a quarter of a century old, and was of limited generalization value because of the uneven socioeconomic distribution amongst Hong Kong's 18 districts, resulting in likely uneven distribution of individual with psychosis amongst them. Other relevant data included data of treated new onset cases from Hong Kong's early intervention service (EASY, annual incidence of at least 600 cases under 25, and estimated 1200-1500 in all age groups), with the limitations of treated incidence discussed above.

The investigators propose a territory-wide epidemiological study of psychosis. The study aims to (1) measure the prevalence of psychotic symptoms in the Hong Kong population; (2) explore associated risk and protective factors for the expression of psychotic symptoms; (3) characterize the functional disability in people with psychotic symptoms; and (4) study the determinant of clinical presentation or non-presentation in people with psychotic symptoms.

ELIGIBILITY:
Inclusion Criteria:

* This study is part of the Hong Kong Mental Morbidity Survey 2010 , the sampling frame is described as follows.

The sample for this survey is planned to represent community dwelling adult population in Hong Kong. The age range will be from 16-75 years. People residing in institutions will not be covered. Only Chinese subjects will be recruited. The survey will adopt a multi-stage sampling design. The sampling frame will consist of a random selection of addresses quarters generated with the help of the Censes and Statistics Department of the Government of Hong Kong SAR. The addresses would be stratified with geographical location and nature of premises. For each address identified, an advance letter with return envelop or contact information will be sent. The advance letter will inform the residents about the nature of the study with an invitation for participation. A maximum of five invitations will be sent by post for non-return within three months. A trained lay interviewer will conduct Phase 1 assessment at home visit for each eligible household expressing interest to participate. To avoid inflation of characteristics that may aggregate within families, only one adult aged 16 years or over will be selected randomly for interview in each household.

Exclusion Criteria:

* The sample frame of the study is described above.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The sample for this survey is planned to represent community dwelling adult population in Hong Kong. The age range will be from 16-75 years. People residing in institutions will not be covered. The survey will adopt a multi-stage sampling design. The sampling frame will consist of a random selection of addresses quarters generated with the help of the Censes and Statistics Department of the Government of Hong Kong SAR. The addresses would be stratified with geographical location and nature of premises. For each address identified, an advance letter with return envelop or contact information will be sent. The advance letter will inform the residents about the nature of the study with an invitation for participation.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2010-08; Primary Completion 2013-08 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Functional Level | Screening
  Social and Occupational Functioning Assessment Scale (SOFAS)

SECONDARY OUTCOMES:
Quality of Life | Screening
  Multidimensional Scale of Perceived Social Support (MSPSS)
Symptomatology | Screening
  Psychosis Screening Questionnaire (PSQ) Beck Scale for Suicide Ideation (BSS) Beck Hopelessness Scale (BHS) Substance Misuse and Dependence Alcohol Use Disorders Identification Test (AUDIT) & Severity of Alcohol Dependence Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: May Mei-ling LAM, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China